CLINICAL TRIAL: NCT01014078
Title: A Four Week Study of Azithromycin Ophthalmic Solution, 1% Versus Placebo in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Mike Schiewe, Associate Director, Inspire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 041-116; P08646
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Azithromycin Ophthalmic Solution, 1% (Experimental)
  Interventions: Drug: Azithromycin Ophthalmic Solution, 1%
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin Ophthalmic Solution, 1% — 1 drop BID for the first 2 days and then 1 drop once a day for the remainder of the study (29 ± 1 days)
  Arms: Azithromycin Ophthalmic Solution, 1%
Drug: Placebo — 1 drop BID for the first 2 days and then 1 drop once a day for the remainder of the study (29 ± 1 days)
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of azithromycin ophthalmic solution, 1% in dry eye subjects over a four week treatment period, using placebo as a comparison.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of dry eye in one or both eyes
* Moderate to severe degree of meibomian gland plugging
* Have best corrected visual acuity in both eyes of at least +0.7 LogMAR
* If female, are non-pregnant or non-lactating

Exclusion Criteria:

* Have anterior blepharitis
* Have lid structural abnormalities
* Have suspected ocular fungal or viral infection
* Have had penetrating intraocular surgery in the past 90 days or require penetrating intraocular surgery during the study
* Have had ocular surface surgery [e.g., laser-assisted in situ keratomileusis (LASIK), refractive, pterygium] within the past year.
* Unable to withhold the use of contact lenses during the study
* Have a known hypersensitivity to azithromycin, erythromycin, any other macrolide antibiotic, or any of the other ingredients in the study medication.
* Have a history of post vitreous detachment.
* Are considered legally blind in 1 eye (LogMAR BCVA= 1.0 or Snellen BCVA= 20/200).
* Have permanent conjunctival goblet cell loss or scarring conditions, including cicatricial blepharitis or conjunctivitis.
* Have a congenitally absent meibomian gland or lacrimal gland.
* Have had cauterization of the punctum or have had punctal plugs (silicone or collagen) inserted or removed within the 90 days prior to the screening.
* Have a serious medical condition which would confound study assessments.
* Have a concomitant ocular pathology that, in the opinion of the investigator, may confound study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Tear Break-Up Time (TBUT) | 4 weeks

SECONDARY OUTCOMES:
Corneal Staining | 4 weeks
Tear Volume | 4 weeks
Meibomian gland plugging | 4 weeks
Subject-rated scores of dry eye symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Chair — Medical Monitor
Locations (9):
- United States (9):
  - Sall Research Medical Center, Inc., Artesia, California
  - David Wirta, MD, Inc., Newport Beach, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Kentucky Lions Eye Center, Louisville, Kentucky
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Abrams Eye Center, Cleveland, Ohio
  - OSU - College of Optometry, Columbus, Ohio
  - Eye Clinics of South Texas, San Antonio, Texas